CLINICAL TRIAL: NCT02724657
Title: THE EFFECTS OF THE BUTEYKO METHOD IN MOUTH BREATHING ASTHMATIC CHILDREN: A CONTROLLED RANDOMIZED STUDY
Brief Title: Buteyko Method for Asthmatic Children With Mouth Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karla Morganna Pereira Pinto de Mendonça, Principal investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.443.588
Record Dates: First submitted 2016-03-07; First posted 2016-03-31 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Asthma; Mouth Breathing
Keywords: Child; Breathing exercises
MeSH Terms: conditions — Asthma; Mouth Breathing

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Buteyko Method (Experimental): Children will perform 6 sessions (twice a week) of treatment with the Buteyko Method.
  Interventions: Other: Buteyko Method
- Control (No Intervention): Asthma education.

INTERVENTIONS:
Other: Buteyko Method — Intervention will be held twice a week during 3 weeks.
  Arms: Buteyko Method

SUMMARY:
To assess the effectiveness of the Buteyko method as an adjunct therapy in the treatment of asthmatic children with mouth breathing.

ELIGIBILITY:
Inclusion Criteria:

* Children from 7 up to 12 years old with asthma diagnose
* Regular inhaled corticosteroids with no change in dose in the preceding 4 weeks.
* Children cannot present: other respiratory disease (such as cystic fibrosis, bronchiectasis, and tuberculosis), retinal detachment, hypertensive crisis, congenital heart defect, pulmonary edema, history of lobectomy or lung segmentectomy, respiratory infections 15 days prior to the evaluations.

Exclusion Criteria:

* Children that are not able to perform some of the necessary procedures, give up participating in the research and present acute symptoms of respiratory tract during the assessments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Sleep disturbance (questionnaire) | Baseline, three weeks later and six months after treatment
  Sleep disturbance will be assessed by the sleep disturbance scale for children (SDSC).

SECONDARY OUTCOMES:
Change in spirometry (FVC, FEV1, FEV1/FVC, FEF25-75%, PEF) | Baseline, three weeks later and six months after treatment
Change in ventilometry (minute volume and vital capacity) | Baseline, three weeks later and six months after treatment
  Minute volume and vital capacity (liters)
Number of hospitalizations | Through study completion, an average of three weeks and six months after treatment
Number of days off-school | During the three weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil